CLINICAL TRIAL: NCT05016570
Title: The Impact of Picture Narrative Format on Knowledge and Acceptability for Lung Screening Print Decision Support Materials
Brief Title: The Impact of Picture Narrative Format on Print Lung Screening Communication Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Katie Robb, Professor of Behavioural Science and Health, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200200021
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Cancer Screening
Keywords: Health Communication; Lung cancer screening; Messages; Comprehension; Visual; Narrative; Comics
MeSH Terms: conditions — Narration

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three groups. They will receive the same lung screening information but the format of this information will be determined by which group they have been randomised to. All participants will complete a questionnaire immediately after viewing the lung screening information.
Who Masked: Investigator
Masking Description: The investigators will be blind to intervention allocation because the intervention and questionnaire is to be undertaken independently and remotely by the participants. Although the intervention is not masked from participants, they will not be informed of the purpose of the study or the different conditions until after they have completed all study measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Picture narrative lung screening information (Experimental): Participants in this arm receive information about lung screening purpose, eligibility, benefits and risks in a format which uses text in combination with sequences of pictures to communicate a coherent message. The designs follow conventions from comics/graphic narratives and key stakeholders were involved during the design process.
  Interventions: Behavioral: Picture narrative information format
- Text with pictures lung screening information (Active Comparator): Participants in this arm receive information about lung screening purpose, eligibility, benefits and risks in a format that uses text with non-narrative pictures for decoration. The pictures have been extracted from the picture narratives being used Arm 1.
  Interventions: Behavioral: Text with pictures information format
- Text-only lung screening information (Active Comparator): Participants in this arm receive information about lung screening purpose, eligibility, benefits and risks in a format that uses text and no pictures.
  Interventions: Behavioral: Text-only information format

INTERVENTIONS:
Behavioral: Picture narrative information format — Lung screening information formatted as picture narratives
  Arms: Picture narrative lung screening information
Behavioral: Text with pictures information format — Lung screening information formatted as text and non-narrative pictures
  Arms: Text with pictures lung screening information
Behavioral: Text-only information format — Lung screening information formatted as text with no pictures
  Arms: Text-only lung screening information

SUMMARY:
The purpose of this study is to test whether a picture narrative format is more successful, than text with pictures or text alone, in communicating lung screening information (primarily defined by positive attitudes towards the design and increase in knowledge) to people likely to be invited to lung screening where available.

DETAILED DESCRIPTION:
Population screening is key to detecting lung cancer early at a more treatable stage. Uptake of screening should be equitable (i.e., screening benefits all eligible members of the population and does not contribute further to health disparities) and informed (i.e., participants have been involved in the decision to take part and their decision aligns with their values and circumstances). Print decision support materials are the primary mechanism for encouraging engagement with cancer screening and supporting decision making. It is essential that we identify print communication techniques that are effective in informing invitees about lung screening.

The intervention, picture narrative information about lung screening, was previously developed through codesign and prototype testing with people likely to be eligible for lung screening (50 to 75 years old, past or current heavy smokers). Participants will be randomised to one of three groups: Picture narrative format, Text with pictures (control 1) or, Text-only (control 2). This study will assess whether presenting lung screening information in a picture narrative format can improve lung cancer screening knowledge, eligibility self-assessment and attitudes. It will also assess whether perceptions of the information designs can explain any impact of the intervention on these outcomes and whether there are differences across socioeconomic groups.

ELIGIBILITY:
Inclusion Criteria:

* Living in Glasgow
* Willing and able to respond unaided to invitation to participate in the trial and give informed consent.
* Aged between 49 and 75 years

Exclusion Criteria:

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Participant Lung Cancer Screening Knowledge scores | Immediately post-intervention
  Participants will be asked 6 multiple choice questions related to the lung screening information presented to the participants during the intervention, covering; Procedure, Eligibility - who, Eligibility - why, Benefits, Adverse effects, Potential results.
Lung Cancer Screening Eligibility self-assessment | Immediately post-intervention
  Concordance between self-reported personal eligibility for lung cancer screening and actual eligibility based on self-reported age and smoking behaviour.
Participant Lung Cancer Screening Attitudes | Immediately post-intervention
  Self-administered four-item lung cancer screening attitudes measure covering cancer fear, fatalism, benefits, and worry, previously used by Smits et al 2018.

SECONDARY OUTCOMES:
Participant Design appraisal ratings | Immediately post-intervention
  Self-administered nine-item measure rating perceptions of appeal, enjoyment, interest, ease of use, trustworthiness, appropriateness, helpfulness, informativity.
  Alongside a single item asking participants whether enough information was provided.

OTHER OUTCOMES:
Treatment compliance | Immediately post-intervention
  Self-reported length of time spent reading the lung screening information.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Robb, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Mental Health and Wellbeing, University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual level study data will be shared via the University of Glasgow's repository Enlighten: Research Data.
Supporting Information: Study Protocol, ICF
Time Frame: On publication of the study results for a period of ten years.
Access Criteria: Data will be made publicly available.